CLINICAL TRIAL: NCT07007780
Title: A Multicenter, Phase II Clinical Study of Sacituzumab Tirumotecan in Neoadjuvant Treatment of Early-Stage TNBC
Brief Title: Sacituzumab Tirumotecan in Neoadjuvant Treatment of Early-Stage TNBC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20252174-F-1
Record Dates: First submitted 2025-05-26; First posted 2025-06-06 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Triple -Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neadjuvant Sacituzumab Tirumotecan (Experimental): Neadjuvant Sacituzumab Tirumotecan
  Interventions: Drug: Sacituzumab Tirumotecan

INTERVENTIONS:
Drug: Sacituzumab Tirumotecan — Sacituzumab Tirumotecan monotherapy before surgery at a dose of 5mg/kg, with a dosing schedule of once every 2 weeks for a total of 12 weeks

SUMMARY:
To explore the application of Sacituzumab Tirumotecan in neoadjuvant treatment of early-stage TNBC, a multicenter, Phase II clinical study of Sacituzumab Tirumotecan in neoadjuvant treatment of early-stage TNBC is proposed. The study aims to evaluate the efficacy and safety of Sacituzumab Tirumotecan and to provide a new treatment option for neoadjuvant treatment of early-stage TNBC.

DETAILED DESCRIPTION:
This study is a multicenter, Phase II clinical trial, planning to enroll 35 eligible early-stage TNBC patients who meet the inclusion and exclusion criteria. Patients will receive neoadjuvant treatment with Sacituzumab Tirumotecan monotherapy before surgery at a dose of 5mg/kg, with a dosing schedule of once every 2 weeks for a total of 12 weeks. Imaging assessments will be conducted every 4 weeks during the neoadjuvant treatment phase. After the neoadjuvant treatment is completed, surgery will be performed within 4 weeks of the last study drug administration. Whether to receive adjuvant treatment after surgery will be determined by the investigator. The primary endpoint of the study is the pathological complete response (pCR) rate. Secondary endpoints include objective response rate (ORR), event-free survival (EFS), overall survival (OS), and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Female subjects aged ≥18 years and ≤70 years at the time of signing the informed consent form.
2. ECOG Performance Status: 0-1.
3. Life Expectancy: Estimated survival of not less than 3 months.
4. Measurable Disease: Presence of at least one measurable lesion according to RECIST 1.1 criteria.
5. Histopathological Diagnosis: Invasive breast cancer, staged as T1c N1-2 or T2-4 N0-2 according to the AJCC classification.
6. TNBC Confirmation: Confirmed as TNBC based on histology and/or cytology, and meeting the following criteria:

   1. HER2-negative: IHC score of 0 or 1+; if IHC is 2+, confirmed negative by fluorescence in situ hybridization (FISH).
   2. ER and PR-negative: IHC showing <1% of cells expressing hormone receptors; in case of multiple pathological results, the molecular subtype of the last biopsy is considered the final subtype.
7. No Prior Systemic Anti-cancer Treatment: No prior systemic anti-cancer treatment.
8. Availability of Tissue Samples: Availability of tissue samples for biomarker testing.
9. Adequate Organ and Marrow Function: (No transfusions, recombinant human thrombopoietin, or colony-stimulating factor within 2 weeks before the first dose), defined as follows:

   1. Hematology: Absolute neutrophil count (NEUT#) ≥1.5×10^9/L; platelets (PLT) ≥100×10^9/L; hemoglobin ≥9 g/dL.
   2. Liver Function: Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) ≤2.5×upper limit of normal (ULN); total bilirubin (TBIL) ≤1.5×ULN.
   3. Renal Function: Creatinine clearance (Ccr) ≥60 ml/min (Cockcroft-Gault formula is provided in the appendix).
   4. Coagulation Function: International normalized ratio (INR), activated partial thromboplastin time (APTT), and prothrombin time (PT) ≤1.5×ULN.
   5. Cardiac Function: Left ventricular ejection fraction (LVEF) ≥50% as shown by echocardiogram (ECHO) or multigated acquisition (MUGA) scan.
10. Contraception: For female subjects of childbearing potential and male subjects with partners of childbearing potential, agreement to use effective medical contraception from the time of signing the informed consent form until 6 months after the last dose.
11. Voluntary Participation: Willingness to participate in the study, signing the informed consent form, having good compliance, and willingness to cooperate with follow-up

Exclusion Criteria:

1. Patients with metastatic breast cancer (Stage IV).
2. Baseline left ventricular ejection fraction (LVEF) <50% as assessed by echocardiogram (ECHO) or multigated acquisition (MUGA) scan at screening, or other significant cardiovascular diseases, or a history of Class III or IV cardiomyopathy described by the New York Heart Association on the same side as the invasive breast cancer.
3. Chemotherapy, endocrine therapy (ET), targeted therapy, and/or radiotherapy for the currently diagnosed breast cancer before enrollment.
4. Previous treatment targeting TROP2 or treatment with a topoisomerase I inhibitor.
5. A history of other malignancies within the past 5 years, excluding cured cervical in situ carcinoma, basal cell carcinoma of the skin, or squamous cell carcinoma of the skin.
6. Known allergy to the study drug or its components.
7. A history of immunodeficiency or organ transplantation.
8. Documented severe dry eye syndrome, severe meibomian gland disease, and/or blepharitis, or a history of corneal diseases that may impede delayed corneal healing.
9. A history of (non-infectious) interstitial lung disease (ILD) or non-infectious pneumonia requiring steroid treatment, current ILD or non-infectious pneumonia, or suspicious ILD or non-infectious pneumonia at screening that cannot be excluded by imaging studies; clinically significant pulmonary impairment due to pulmonary comorbidities, including but not limited to any underlying pulmonary disease (e.g., pulmonary embolism within 3 months before dosing, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion, etc.) or any autoimmune, connective tissue, or inflammatory diseases that may involve the lungs (e.g., rheumatoid arthritis, Sjögren's syndrome, sarcoidosis, etc.), or a history of pneumonectomy.
10. Active autoimmune disease requiring systemic treatment within the past 2 years (hormone replacement therapy is not considered systemic treatment, such as Type I diabetes, hypothyroidism requiring only thyroid hormone replacement, adrenal or pituitary insufficiency requiring only physiologic doses of glucocorticoid replacement).
11. Active infection requiring systemic treatment within 2 weeks before the first dose.
12. Any comorbidities that, in the investigator's judgment, pose a serious risk to patient safety or may affect the patient's ability to complete the study, including but not limited to uncontrolled hypertension, severe diabetes, active infections, etc.
13. Any condition or other circumstances that the investigator believes may interfere with the evaluation of the study drug, the safety of the subject, or the interpretation of the study results, or any other condition that the investigator deems unsuitable for participation in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | At the end of Cycle 1 (each cycle is 14 days)

SECONDARY OUTCOMES:
adverse effects | through each neoadjuvant chemotherapy Cycle (each cycle is 14 days)]
  Serious adverse effect occur within neoadjuvant chemotherapy
Objective Reaponse Rate(ORR) | At the end of every cycle (each cycle is 14 days)
Event-free survival (EFS) | Up to 2 years
  Defined as the time from treatment initiation to the first occurrence of any of the following events: disease progression precluding surgical treatment, local or distant recurrence, or death from any cause.